CLINICAL TRIAL: NCT00326534
Title: Rickettsial Genesis to Sarcoidosis in Denmark
Status: Completed | Type: Observational
Sponsor: Statens Serum Institut (Other)
Collaborators: Bispebjerg Hospital (Other); Civilingeniør Johs. E. Ormstrup og Hustru Grete Ormstrups Fond (Unknown)
Responsible Party: Claus Bo Svendsen, MD, Statens Serum Institut
Other Study IDs: KF 01 303797; 2006-41-6575
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Sarcoidosis; Rickettsia Infections
Keywords: Sarcoidosis; Rickettsia; Serological reactions; Polymerase chain reaction
MeSH Terms: conditions — Sarcoidosis; Rickettsia Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coats, serum, bronchoalveolar lavage fluid and transbronchial biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Patients without sarcoidosis, but requiring a fiberoptic bronchoscopy
- Sarcoidosis patients: Patients with newly diagnosed sarcoidosis

SUMMARY:
One study has suggested a connection between an infection with Rickettsia species and sarcoidosis finding molecular evidence of rickettsial deoxyribonucleic acid (DNA) in two patients. Another study found no antibodies in twenty Swedish patients with sarcoidosis.

This study will further enhance the subject by three different approaches in Danish patients.

The purpose of this study is to find serological and molecular evidence of an infection with Rickettsia species in Danish patients with sarcoidosis.

DETAILED DESCRIPTION:
The study has three approaches to the subject:

1. A serological survey of rickettsial immunoglobin G (IgG)-antibodies in 50 patients with sarcoidosis compared to 50 blood donors without sarcoidosis.
2. An archival study using pre-existing lymph node biopsies, where immunohistochemical analysis, fluorescent in situ hybridization, and polymerase chain reaction will be applied to samples from 50 patients with sarcoidosis and compared to 50 patients without sarcoidosis and 10 patients with tuberculosis.
3. A prospective study using bronchoscopically obtained samples from 20 patients with sarcoidosis, compared to 20 patients without sarcoidosis. The study applies the same techniques as the second study, but enhancing the information from the patients.

ELIGIBILITY:
Inclusion Criteria:

* Referred to fiberoptic bronchoscopy in the department either because of sarcoidosis, hemoptysis, chronic cough, or cancer suspicion

Exclusion Criteria:

* Pregnant patients
* Patients under the age of 18
* Patients without consent
* Patients with a registered wish of not having their samples used for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to fiberoptic bronchoscopy in the department either because of sarcoidosis, hemoptysis, chronic cough, or cancer suspicion
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Svendsen, MD, Principal Investigator — Statens Serum Institut; Nils Milman, MD, Study Chair — Rigshospitalet, Denmark; Karen A Krogfelt, PhD, Study Chair — Statens Serum Institut
Locations (1):
- Denmark, Copenhagen S, Denmark

REFERENCES:
- [Background] Planck A, Eklund A, Grunewald J, Vene S. No serological evidence of Rickettsia helvetica infection in Scandinavian sarcoidosis patients. Eur Respir J. 2004 Nov;24(5):811-3. doi: 10.1183/09031936.04.00014604. PMID 15516677
- [Background] Nilsson K, Pahlson C, Lukinius A, Eriksson L, Nilsson L, Lindquist O. Presence of Rickettsia helvetica in granulomatous tissue from patients with sarcoidosis. J Infect Dis. 2002 Apr 15;185(8):1128-38. doi: 10.1086/339962. Epub 2002 Mar 21. PMID 11930323
- [Result] Svendsen CB, Milman N, Hoier-Madsen M, Dziegiel MH, Krogfelt KA. Determination of rickettsial and antinuclear antibodies in Danish patients with sarcoidosis. Clin Respir J. 2008 Oct;2(4):202-7. doi: 10.1111/j.1752-699X.2008.00051.x. PMID 20298335